CLINICAL TRIAL: NCT06666400
Title: Living Healthy for Moms (LHM) Randomized Type I Hybrid EffectivenessImplementation Trial: A Doula-Delivered Cognitive Behavioral Training (CBT) + Cardiovascular Health (CVH) Intervention for Birthing Individuals
Brief Title: Living Healthy for Moms RCT
Acronym: LHMoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Weill Medical College of Cornell University (Other); Northern Manhattan Perinatal Partnership (Other); New York City Health and Hospitals Corporation (Other); Caribbean Women's Health Association (Unknown)
Responsible Party: Principal Investigator, Mary E. D'Alton, Chair of the Department of Obstetrics and Gynecology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAV1436; 5U54HD113172-02 (NIH)
Record Dates: First submitted 2024-10-17; First posted 2024-10-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD); Cardiac Event
Keywords: severe maternal morbidity; maternal mortality; mental health; cardiovascular events; health disparity; maternal welfare; structural racism
MeSH Terms: conditions — Depression, Postpartum; Cardiovascular Diseases; Maternal Death; Psychological Well-Being; Systemic Racism

STUDY DESIGN:
Intervention Model Description: This randomized type 1 Hybrid Effectiveness-Implementation Trial will enroll 600 birthing individuals post-delivery, while they are still in the hospital, pre-discharge. These individuals will be randomized to one of two groups: the LHM arm (N=300) will receive a CBT+ Cardiovascular Health (CVH) Intervention to reduce CV risk, and the attention control arm (N=300) will receive standard doula care and the same number of telephone or video call-delivered sessions on general health education topics not related to CV health or depression.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (Active Comparator): The attention control arm (N=300) will receive standard doula care and the same number of telephone or video-delivered sessions and will last the same amount of time on general postpartum health topics not related to CV health or depression. Attention control participants will not receive doula-initiated outreach during the first 7 days.
  Interventions: Other: No intervention
- LHMoms Intervention Arm (Experimental): The LHM arm (N=300) will receive a CBT+ Cardiovascular Health (CVH) Intervention to reduce CV risk. LHM employs a cognitive behavioral training (CBT) + cardiovascular health (CVH) intervention delivered by doulas and integrating a healthy lifestyle intervention to reduce CV risk. The LHM intervention integrates the following key elements: (1) doula-led emergency detection in the first 7 days post-discharge; (2) home BP monitoring (HBPM); and (3) 11-sessions of the doula-delivered intervention to prevent PPD and reduce CV risk from 1 week to 6 months post-discharge, supported by (4) education through the Patient-Activated Learning System (PALS), a novel education platform used to engage low-literacy, racially marginalized individuals. LHM is based on the Thinking Healthy Programme (THP), an intervention originally designed to treat PPD in low and middle-income countries using community health workers.
  Interventions: Behavioral: LHMoms Intervention

INTERVENTIONS:
Behavioral: LHMoms Intervention — The LHM arm (N=300) will receive a CBT+ Cardiovascular Health (CVH) Intervention to reduce CV risk. LHM employs a (CBT) + cardiovascular health (CVH) intervention delivered by doulas and integrating a healthy lifestyle intervention to reduce CV risk. The LHM intervention integrates the following key elements: (1) doula-led emergency detection in the first 7 days post-discharge; (2) home BP monitoring (HBPM); and (3) 12-sessions of the doula-delivered intervention to prevent PPD and reduce CV risk from 1 week to 6 months post-discharge, supported by (4) education through the Patient-Activated Learning System (PALS), a novel education platform used to engage low-literacy, racially marginalized individuals. LHM is based on the Thinking Healthy Programme (THP), an intervention originally designed to treat PPD in low and middle-income countries using community health workers.
  Other Names: LHM Arm
  Arms: LHMoms Intervention Arm
Other: No intervention — Standard doula care and the same number of telephone or video-delivered sessions and will last the same amount of time on general postpartum health topics not related to CV health or depression. Attention control participants will not receive doula-initiated outreach during the first 7 days.
  Arms: Attention Control

SUMMARY:
LHMoms is a novel integrated care intervention that focuses intensively on care continuity and community-to-healthcare linkages for postpartum birthing individuals. The intervention starts prior to discharge in the delivery hospitalization and extends to six months post-partum, thus covering critical windows to prevent long-term physical and mental health sequelae.

DETAILED DESCRIPTION:
Most preventable maternal deaths occur in the intrapartum and immediate postpartum (PP) periods, as do complications from undetected/undertreated mental health (MH) conditions (e.g., suicide, overdose) and cardiovascular (CV) events. In New York City (NYC), maternal deaths are 8-12 times higher for Black than for White birthing parents. However, most community-based programs addressing the health of birthing individuals in this population have been narrowly focused on basic services (e.g., breastfeeding, social support), with limited focus on evidence-based care. Holistic interventions addressing physical, mental, and social health needs in the critical PP transition and moving from trauma- and "risk"-based to a strength- and empowerment-based approach are urgently needed. Many hospital, community, and governmental barriers preclude broad adoption and scaling of doula-delivered care, and it is not known how facilitators, assets, and resources can improve care continuity and community-hospital linkages to support birthing individuals at diverse sites across NYC. The impact of doula-led interventions at patient- and health-system levels have yet to be rigorously evaluated. In collaboration with the Caribbean Women's Health Association and the Northern Manhattan Perinatal Partnership, this study will address these gaps by implementing and evaluating Living Healthy for Moms (LHMoms) in three complementary settings and populations (Brooklyn, Queens, and Northern Manhattan). LHMoms is a novel integrated care intervention that focuses intensively on care continuity and community-to-healthcare linkages that starts prior to discharge and during the first 7 days post-discharge (PD) and extends into six months post-partum, as critical windows to prevent long-term physical and mental health sequelae, while also addressing key determinants of lifelong health risk. The investigators have developed several innovative, evidence-based interventions, including an online education empowerment program (using a Patient Activated Learning System platform we developed) to build patient self-advocacy beginning in-hospital; a doula-led health emergency detection program during the critical first 7 days PD; and a trauma-informed doula-delivered cognitive behavioral training (CBT) intervention to address PP depression and cardiovascular risks for the critical six months following delivery. This study proposes a rigorous, mixed-methods study of LHMoms to address three specific aims. In Aim 1, the study will test the effectiveness of LHMoms vs. attention control in a Hybrid Type 1 Implementation Trial with 600 randomized birthing individuals at three hospital sites in Brooklyn, Queens, and Northern Manhattan. This will include refining and tailoring the intervention to each site to maximize care quality, building capacity for doulas to deliver LHMoms, and assessing effectiveness in lowering PP depression, improving CV health. In Aim 2, the study will analyze the effects of LHMoms on PP healthcare utilization and satisfaction. In Aim 3, the study will examine the implementation process and outcomes of the LHMoms intervention at the three sites. This project will advance the overall goals of NY-CHAMP to optimize PP outcomes for historically disadvantaged birthing individuals.

ELIGIBILITY:
Inclusion Criteria:

* Birthing individuals aged 18 years or older
* Delivery of singleton live birth; and
* Minority race (self-identified Black), minority ethnicity (self-identified Latinx), and/or Medicaid beneficiary.

Exclusion Criteria:

* Individuals unable to conduct visits and complete surveys via computer or phone,
* Younger than 18 years
* Individuals unable to communicate (reading, writing, speaking) in English, Spanish or Haitian Creole
* multifetal pregnancy
* gestational age less than 24 weeks at delivery
* known major fetal anomaly in current pregnancy
* known fetal demise
* on hemodialysis
* active user of IV drugs
* active suicidal ideation with intent and plan
* known primary psychotic disorder
* plans to move out of the area within 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) score | 6 months post hospital discharge
  The primary outcome of PPD, operationalized as the presence or absence of postpartum depressive symptoms, is defined by EPDS score (≥9). EPDS ≥9 was chosen specifically because that is the score used as the cut-off to refer for clinical evaluation, and the rate of EPDS ≥9 ranges from about 30-40% depending on other characteristics of the clinics. Assuming 1:1 randomization, a design effect of 1.5 to account for variance among sites and doulas, a power of 0.80, a two-sided significance level of 0.05, and 20-25% attrition, to detect a PPD symptom rate reduction from 33.5% in the control arm to 23% in the intervention, a sample size of approximately 450 individuals (225 in each study arm) is needed. The EPDS scale ranges from 0 to 30, and a higher score indicates more severe depression.
Heart Score | 6 months post hospital discharge
  The "Heart Score" is a metric calculated through the American Heart Association's online calculator. It incorporates the behavioral and biological components Life's Essential 8 (LE8) (diet, physical activity, nicotine exposure, sleep health, body mass index, blood lipids, blood glucose, and blood pressure). These components will be collected from participants during the study but are not being assessed as individual outcomes; instead, the Heart Score from 1-100 as calculated by the AHA online calculator will be used as the outcome of CV health.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. D'Alton, MD, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York City Health + Hospitals/ Queens, Jamaica, New York
  - NewYork-Presbyterian Allen Hospital, New York, New York
  - Weill Cornell Medicine, New York, New York

REFERENCES:
- [Derived] Faiz JM, Bylinsky I, Rincones Rojas L, Kopatsis K, St Clair V, Dorval-Moller M, Voegtline K, Lipkind H, Safford MM, Hall KS, Reddy U, Osborne LM. Doula-Delivered Cognitive Behavioral Training and Cardiovascular Health Intervention for Birthing Individuals in a Low-Income New York City Population: Protocol for a Living Healthy for Moms Randomized Type I Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2025 Dec 10;14:e76871. doi: 10.2196/76871. PMID 41370009